CLINICAL TRIAL: NCT05680090
Title: Prospective Validation of an Artificial Intelligent System for Eye Emergency Triage and Primary Diagnosis
Brief Title: Artificial Intelligent System for Eye Emergency Triage and Primary Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Other Study IDs: 2021KYPJ046
Record Dates: First submitted 2022-12-13; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Emergencies; Eye Diseases
Keywords: Artificial intelligence; Ophthalmic emergency triage; Primary diagnosis; Multimodal data
MeSH Terms: conditions — Emergencies; Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eligible participants for AI-based ophthalmic emergency triage and primary diagnosis
  Interventions: Diagnostic Test: Artificial intelligent system for eye emergency triage and primary diagnosis

INTERVENTIONS:
Diagnostic Test: Artificial intelligent system for eye emergency triage and primary diagnosis — An intelligent triage and diagnostic system for ophthalmic emergencies has been developed. In the prospective test, patients with acute ocular symptoms can achieve remote self-triage and primary diagnosis after uploading metadata and ocular images.

SUMMARY:
Ophthalmic emergencies are acute vision-threatening disorders, for which a delay in prompt emergency response could result in catastrophic vision loss. Triage is an effective process for ensuring that timely emergency care is provided despite limited resource by prioritizing patients to appropriate orders for visits. Historically, registered nurses classify emergency patients based on personal experiences with high variation. Additionally, primary healthcare providers have been conventionally at the forefront of providing first aid care. However, most of ocular emergencies are wrongly diagnosed or referred due to non-eye specialists' limited knowledge and training in the ophthalmology.

Here, the investigators established and validated an artificial intelligence system, EE-Explorer, to triage eye emergencies and assist in primary diagnosis using metadata and ocular images. This system has been integrated into a website to be prospectively validated in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Suffering acute ophthalmic symptoms within one month
2. Visiting the ocular emergency department for the first time
3. Must be able to complete the triage form for ophthalmic emergency
4. Must be able to cooperate either by submitting smartphone photographs or receiving slit-lamp examination

Exclusion Criteria:

The image quality does not meet the clinical requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Through the online popular science, news reports, and other channels, we will promote and inform patients about the relevant knowledge of ophthalmic emergencies, so that they can judge by themselves and freely decide whether to participate in this study or not.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-01-13 (Estimated); Study Completion 2023-01-20 (Estimated)

PRIMARY OUTCOMES:
The accuracy of the triage model | 2023.1
  Use the triage model to classify patients with acute ocular symptoms, and count the proportion of correct classification.

SECONDARY OUTCOMES:
The accuracy of the primary diagnostic model | 2023.1
  Use the primary diagnostic model to diagnose patients with ophthalmic emergencies, and count the proportion of correct diagnosis in all patients.

OTHER OUTCOMES:
Acceptance of the patients | 2023.1
  Questionnaire scores

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China